CLINICAL TRIAL: NCT07286071
Title: Safety and Efficacy of Using Traditional Ureteral Access Sheath Versus Flexible and Navigable Suction Sheath in Retrograde Intra-Renal Stone Surgery for Renal Stones ≤ 20 mm: A Randomized Controlled Study
Brief Title: Safety and Efficacy of Traditional Versus Flexible and Navigable Suction Sheath in Retrograde Intra-Renal Stone Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hassan mahmoud hassan, Resident of Urology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU_MS401_2025
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Urolithiasis; Kidney Calculi; Nephrolithiasis
Keywords: Urolithiasis; Kidney Calculi; RIRS; UAS; Suction UAS; Endourology; Laser Lithotripsy; Stone-Free Rate
MeSH Terms: conditions — Urolithiasis; Kidney Calculi; Nephrolithiasis | interventions — Suction

STUDY DESIGN:
Intervention Model Description: Two groups of participants were assigned in parallel. One group underwent retrograde intrarenal surgery using a ureteral access sheath with suction. The other group underwent retrograde intrarenal surgery using a traditional ureteral access sheath without suction. Both groups were followed to compare safety and effectiveness outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suction Ureteral Access Sheath Group (Experimental): Participants in this group underwent retrograde intrarenal surgery using a ureteral access sheath equipped with a suction mechanism. After anesthesia, a guide wire was placed and the ureter was evaluated. The suction ureteral access sheath was inserted over the guide wire and positioned inside the kidney near the stone. Controlled negative pressure was applied to improve removal of stone fragments and to maintain lower pressure inside the kidney during the procedure. Laser lithotripsy was performed, and stone fragments were aspirated through the suction system. A double-J ureteral stent was placed at the end of the procedure.
  Interventions: Procedure: Retrograde intrarenal surgery using a ureteral access sheath with suction
- Traditional Ureteral Access Sheath Group (Active Comparator): Participants in this group underwent retrograde intrarenal surgery using a traditional ureteral access sheath without suction. After anesthesia and guide wire placement, the traditional ureteral access sheath was inserted and positioned below the junction between the ureter and the kidney. Laser lithotripsy was performed in the standard manner. Stone fragments were removed passively using irrigation and by repeatedly retrieving fragments with a basket. A double-J ureteral stent was placed at the end of the procedure.
  Interventions: Procedure: Retrograde intrarenal surgery using a traditional ureteral access sheath

INTERVENTIONS:
Procedure: Retrograde intrarenal surgery using a ureteral access sheath with suction — This intervention involves performing retrograde intrarenal surgery using a ureteral access sheath equipped with a suction mechanism that applies controlled negative pressure to help remove stone fragments and manage pressure inside the kidney during the procedure.
  Arms: Suction Ureteral Access Sheath Group
Procedure: Retrograde intrarenal surgery using a traditional ureteral access sheath — This intervention involves performing retrograde intrarenal surgery using a conventional ureteral access sheath without suction, relying on irrigation flow and basket retrieval for stone fragment removal.
  Arms: Traditional Ureteral Access Sheath Group

SUMMARY:
This study compares two techniques used during RIRS for the treatment of kidney stones measuring up to 20 mm. During RIRS, surgeons often use a device called a UAS to help pass instruments into the urinary system and to assist with the removal of stone fragments. A traditional UAS allows irrigation fluid and small fragments to flow out passively. A newer type, known as a suction UAS, applies controlled negative pressure to help clear stone fragments more effectively and may reduce pressure inside the kidney during the procedure.

The purpose of this study is to determine whether the suction UAS offers better clinical outcomes than the traditional UAS. The main outcomes assessed include the SFR, the duration of surgery, and complications after the procedure such as fever, sepsis, urinary infection, calyceal injury, or ureteral injury.

In this randomized study, adult patients undergoing RIRS for a single renal stone were assigned to either the suction UAS or the traditional UAS. All patients were followed after surgery to assess stone clearance and any complications. The results of this study aim to provide evidence on whether suction UAS improves safety or effectiveness in RIRS compared with the traditional approach.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged eighteen years or older
* Male or female participants
* Presence of a single kidney stone measuring up to twenty millimeters
* Candidate for retrograde intrarenal surgery according to clinical evaluation
* Able and willing to provide informed consent

Exclusion Criteria:

* Active or untreated urinary infection
* History of open kidney surgery or kidney trauma
* Contraindications to anesthesia, including uncontrolled diabetes, severe cardiac disease, or significant coagulation disorders
* Presence of ureteral narrowing or obstruction at the junction between the ureter and the kidney
* Positive urine culture that does not resolve after appropriate treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Stone-free rate | One month after surgery
  The stone-free rate represents the proportion of participants who show no residual stone fragments or only clinically insignificant small fragments on postoperative imaging. Imaging is performed using non-contrast computed tomography. Findings are classified into four categories based on fragment size: complete clearance, fragments up to two millimeters, fragments between two point one and four millimeters, and fragments larger than four millimeters. The outcome is expressed as the percentage of participants achieving complete clearance or clinically insignificant fragments.

SECONDARY OUTCOMES:
Duration of surgery | During surgery
  Total time required to complete the surgical procedure, measured from the insertion of the ureteroscope until placement of the ureteral stent.
Readmission after surgery | Within one month after surgery
  Number of participants requiring hospital readmission for pain, infection, or any complication related to the surgery.
Need for an additional procedure | Within three months after surgery
  Proportion of participants requiring a second surgical intervention to remove remaining stone material.
Urinary infection after surgery | Within one month after surgery
  Occurrence of laboratory-confirmed urinary infection requiring medical treatment, classified using the Clavien-Dindo system.
Systemic infection after surgery | Within one month after surgery
  Occurrence of systemic infection requiring medical intervention, including antibiotic therapy or hospitalization, assessed using the Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Department of Urology, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the study will be made available after removal of all direct identifiers. The shared data will include demographic information, clinical characteristics, surgical details, and outcome measurements related to stone clearance and postoperative events. Data will be provided only for the purpose of scientific research and verification of study findings.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available starting six months after publication of the main study results. The data will remain accessible for a period of five years from the date of release.
Access Criteria: Researchers who wish to access the data must submit a written request that includes a summary of the research objectives and the intended use of the data. Approval will require review by the study investigators. Upon approval, data will be shared through a secure data transfer method. Recipients must agree not to attempt to reidentify participants and must use the data only for the approved research purpose.